CLINICAL TRIAL: NCT04767256
Title: Intravenous Dexamethasone and Dexmedetomidine on the Analgesic Efficacy of Erector Spinae Plane Block for Posterior Lumbar Interbody Fusion Surgery
Brief Title: Intravenous Dexamethasone and Dexmedetomidine on the Analgesic Efficacy of Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xi Wu, Principal Investigator, Department of Anesthesiology, Union Hospital of Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH20210202
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Dexamethasone; Dexmedetomidine; Nerve Block
MeSH Terms: interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DD group (Experimental): co-administered intravenous dexamethasone 10 mg and dexmedetomidine 1 ug/kg
  Interventions: Drug: Dexamethasone and dexmedetomidine; Other: Ultrasound-guided lumbar erector spinae plane block; Other: PCIA
- D group (Placebo Comparator): intravenous dexmedetomidine 1 ug/kg
  Interventions: Drug: Dexmedetomidine; Other: Ultrasound-guided lumbar erector spinae plane block; Other: PCIA

INTERVENTIONS:
Drug: Dexamethasone and dexmedetomidine — General anesthesia was induced with sufentanil 0.5-0.8 ug/kg, propofol 1.5-2.0 mg/kg, and rocuronium 0.5-1.0 mg/kg. Intravenous dexamethasone 10 mg was injected and a 50-ml syringe containing dexmedetomidine 1 ug/kg in 0.9% saline was infused after induction of general anaesthesia over a 30-min period. Anesthesia was maintained by remifentanil and sevoflurane to keep the Narcotrend index reading between 40 and 60.
  Arms: DD group
Drug: Dexmedetomidine — Intravenous dexmedetomidine 1 ug/kg was infused after induction of general anaesthesia over a 30-min period.
  Arms: D group
Other: Ultrasound-guided lumbar erector spinae plane block — The probe was installed in the sagittal axis in the midline at the L3 vertebral level. The spinous processes were ﬁrst visualized, after which the probe was lateralized, and the transverse processes and the erector spinae muscle were visualized approximately 3 cm laterally to the midline. The needle was advanced between the transverse process and the deep fascia of the erector spinae muscle from the caudal to the cranial using in-plane technique. The location of the needle was confirmed with 2mL saline solution, after which 20 mL of 0.4% ropivacaine was administered.
Other: PCIA — Intravenous PCA included 0.9% saline with sufentanil and was programmed to run at 2ml with a 1-ml bolus dose and a 10-min lockout time. The patients with VAS more than 4 despite using intravenous PCA were treated with rescue analgesics comprising intravenous parecoxib.

SUMMARY:
Patients having lumbar spinal fusion often complain about severe postoperative pain and postoperative rehabilitation process can be affected negatively. Postoperative pain that cannot be well controlled may lead to delayed mobilization, pulmonary and thromboembolic complications, prolonged hospital stays, and chronic pain syndromes. Pain after spinal surgery can arise from several different tissues, such as the vertebrae, disks, ligaments, dura, facet joint, muscle, fascia, and subcutaneous and cutaneous tissues.

Ultrasound-guided lumbar erector spinae plane block (ESPB) has been shown to reduce postoperative pain in patients undergoing posterior lumbar interbody fusion (PLIF). However, the duration of analgesia after single-shot ESPB with commonly used local anesthetics is reported to be no more than 12 h, which often not long enough to provide satisfactory postoperative pain relief, as the pain typically lasts for several days. Compared with perineural route, intravenous additives to local anesthetics are commonly accepted as its safety and efficiency have been reported. Moreover, co-administration of intravenous dexamethasone and dexmedetomidine significantly prolonged the time to ﬁrst rescue analgesic request after single-shot interscalene brachial plexus block. However, more data are needed especially for lumbar ESPB.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 yrs
2. American Society of Anesthesiologists physical statusⅠ-Ⅲ
3. Involvement of ≤3 spinal levels
4. Undergo elective posterior lumbar interbody fusion
5. Informed consent

Exclusion Criteria:

1. A known allergy to the drugs being used
2. Pre-existing neuropsychiatric disorders or language barrier
3. Analgesics intake, history of substance abuse
4. Contraindications to peripheral nerve block
5. Acute cerebrovascular disease
6. Severe liver failure
7. Uncontrolled low blood pressure
8. Sinus bradycardia or atrioventricular block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The cumulative opioid consumption | At 24 postoperative hours
The time to ﬁrst rescue analgesic request | Up to 48 postoperative hrs

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 6, 12, 18, 24, 30, 36, 42, and 48 hrs after the surgery
Incidence of postoperative nausea and vomiting | Up to 24 postoperative hrs
Postoperative hospital length of stay | Up to 3 weeks
Adverse events | Up to 48 postoperative hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No